CLINICAL TRIAL: NCT05794412
Title: Mucosal Immunity: Influence on Infectious Viral Load: a Prospective Observational Study
Acronym: MIViral
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other); ModernaTX, Inc. (Industry)
Responsible Party: Principal Investigator, Isabella Eckerle, Prof., University Hospital, Geneva
Other Study IDs: 2022-01722
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: SARS-CoV-2 Infection; Influenza Viral Infections; Virus Shedding; Mucosal Immunity; RSV Infection
MeSH Terms: conditions — COVID-19; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to learn about the influence of pre-existing mucosal immunity, i.e. antibodies and immune cells that are present at the nasal mucosa before infection, on the infectious viral load after infection with SARS-CoV-2, influenza virus and RSV. The investigators will include app. 320 participants which will be followed for up to 17 months. During this time, the investigators will monitor their nasal mucosal antibodies at regular intervals and compare them to their infectious viral load if they are infected with SARS-CoV-2, influenza virus or RSV. Participants are invited to take a test for SARS-CoV-2, influenza virus or RSV in case of respiratory symptoms. If participants are positive the investigators will follow their viral load kinetics by taking nasopharyngeal swabs every 2-3 days. The investigators will also record the duration and strength of the following symptoms:

* Cough
* Fever
* Tired
* Sore throat
* Difficulty breathing
* Respiratory distress
* Headache
* Loss (or alteration) of smell
* Loss (or alteration) of sense of taste
* Myalgias
* Chills
* Subjective fever
* Pink sputum (or coughing up blood)
* Thoracic pain
* Runny nose
* Abdominal pain
* Nausea
* Vomiting
* Diarrhea
* Constipation
* Irritated or watery eyes
* Rashes
* Other

ELIGIBILITY:
Inclusion Criteria:

* In general good health, as determined by study investigators
* All participants must be living in the canton of Geneva or working/studying in the canton of Geneva and living in neighboring communities that are within one hour travelling distance by car.

Exclusion Criteria:

* Inability to provide written consent.
* Severely immunocompromised subjects as determined by the study investigator
* Treated with inhaled drugs by nasal route within the last month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infectious viral load | up to 14 days post symptom onset

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Meyer, Dr., Principal Investigator — University of Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided